CLINICAL TRIAL: NCT07111676
Title: Evaluating the Efficacy and Cost-effectiveness of the School-based Solution-focused Intervention for Mental Health (SIM) in First Year of Upper Secondary School Students
Brief Title: Evaluation of the School-based SIM Program in Upper Secondary School Students
Acronym: SIMRCT1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 284745; 2023-00581_3 (Other Grant/Funding Number: Swedish Research Council for Health, Working Life and Welfare); OLL-1022722 (Other Grant/Funding Number: The Foundation for Medical Research at Örebro University Hospital - Nyckelfonden)
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Solution-focused Capability; Mental Well-being; Mental Problems; Perceived Stress
Keywords: Mental well-being; Solution-focused Intervention for mental health; SIM; School-based intervention; Strength-based; Mental health promotion; Solution-focused coaching; Cluster randomized controlled trial; Adolescents; Solution-focused brief therapy; Universal mental health intervention
MeSH Terms: conditions — Psychological Well-Being | interventions — Mental Health

STUDY DESIGN:
Intervention Model Description: A two-arm, cluster, randomized controlled trial is conducted with an intervention group receiving SIM and a control group receiving a lecture on mental well-being along with usual school provision. Randomization is done by class as the intervention takes place in mentor groups. Based on the results of the largest of our feasibility studies, paired measurements on 559 students are required to detect a small effect in mental well-being with 80% power (d=0.196) and a significance level of 0.05. The evaluation is based on validated instruments and measurements before and after the intervention and after 6 and 9 months. To answer the primary research question, we will analyze the mean difference in mental well-being between the intervention and control groups using a linear mixed effects regression model with a random effect for school class. Variables identified as important predictors of the outcome will be included in the regression model in order to reduce outcome variance.
Masking Description: Masking of conditions for the students will be used up until consent and baseline measures have been completed. After that, masking in this evaluation is not practically possible.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Students participating in the school-based SIM program designed to promote mental well-being.
  Interventions: Behavioral: The Solution-focused Intervention for Mental health (SIM)
- Control group (No Intervention): Students receiving a lecture on mental well-being along with usual student health provision.

INTERVENTIONS:
Behavioral: The Solution-focused Intervention for Mental health (SIM) — SIM is a manual-based program delivered to upper secondary school students in mentor groups by a specially trained teacher. It consists of group-based, solution-focused coaching set within a normative frame of mental well-being. By co-creating perceptions and meaning through language and dialogue, focusing on resources for approaching a preferred future, students increase their solution-building capability, thereby acquiring skills to become agents in their own life, more aware of and prone to invest in mental health. For a detailed description, see Söderqvist et al. https://doi.org/10.1016/j.ssmmh.2025.100493.
  Arms: Intervention group

SUMMARY:
Söderqvist et al. recently reported on a new school-based program designed to promote mental well-being in adolescents: the Solution-Focused Intervention for Mental Health (SIM, https://doi.org/10.1016/j.ssmmh.2025.100493). While previous studies on SIM were designed mainly to test, develop, refine and improve the program and its feasibility in a school setting, the current project aims to test the efficacy of SIM on adolescent mental health, primarily mental well-being.

A two-arm, cluster, randomized, controlled trial will be conducted. The intervention group will receive the SIM program, and the control group will receive a lecture on mental well-being along with the usual school provisions. Randomization is done by class because the intervention takes place in mentor groups. Based on the results of our largest feasibility study, 559 students are required for paired measurements to detect a small effect on mental well-being with 80% power and a significance level of 0.05. The evaluation is based on validated instruments, with measurements taken before and after the intervention, as well as six and nine months later. The project is being implemented in collaboration with six upper secondary schools in Sweden. Recruitment and anchoring at the participating schools, as well as class randomization strafied on educational program, took place in 2025. Enrollment of participating students will begin in January 2026.

This project will contribute new knowledge to the field by evaluating a universal program for schools to use in their health promotion work. The latter is important since high levels of mental well-being independently predict a lower incidence of subsequent mental illness and have a range of positive effects on individuals and society.

ELIGIBILITY:
Inclusion Criteria:

* first and second-year upper secondary school students
* students enrolled in regular school programs

Exclusion Criteria:

* students with insufficient knowledge of the Swedish language
* students who are absent during the information meeting or could not be reached for a separate meeting to receive the accurate information
* students who are absent at the start session or cannot be reached to complete the baseline prior to the first themed SIM session
* students who for various reasons (e.g. functional impairments) are unable to participate in an ordinary teaching situation.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Mental well-being | This study will examine participants from enrollment to the end of the 10-week intervention, as well as at six- and nine-month follow-ups.
  The mean difference in mental well-being between the intervention and control arms as measured by the Mental Health Continuum - Short Form. For more on the measurement instrument, see Söderqvist and Larm, https://doi.org/10.1007/s12144-021-01626-6.

SECONDARY OUTCOMES:
Mental problems | This study will examine participants from enrollment to the end of the 10-week intervention, as well as at six- and nine-month follow-ups.
  The difference in mental problems between the intervention and control arms as measured by the Revised Child Anxiety and Depression Scale 25. For more on the measurement instrument, see Carlander et al. https://doi.org/10.1002/mpr.2007.
Perceived stress | This study will examine participants from enrollment to the end of the 10-week intervention, as well as at six- and nine-month follow-ups.
  The difference in perceived stress between the intervention and control arms as measured by a 14-item scale comprising stressors associated with different areas of adolescent life.

OTHER OUTCOMES:
Solution-building Capability | This study will examine participants from enrollment to the end of the 10-week intervention, as well as at six- and nine-month follow-ups.
  The difference in solution-building capability between the intervention and control arms as measured by a modified 15-item version of the Solution Building Inventory originally developed by Grant et al (2012).

IPD SHARING:
Plan to Share IPD: Undecided
Data can be made available by the authors upon reasonable request, for researchers who meet the criteria for access to confidential data. At this point, a decision to publicly share data cannot be made because of ethical and legal restrictions concerning the student's consent and data ownership. The data will be owned by a third party, which have imposed restrictions.